CLINICAL TRIAL: NCT01383174
Title: Nuevo Amanecer: Promoting the Psychosocial Health of Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: California Breast Cancer Research Program (Other); Circulo de Vida Cancer Support and Resource Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15BB-1300; 15BB-1301 (Other Grant/Funding Number: California Breast Cancer Research Program)
Record Dates: First submitted 2011-06-03; First posted 2011-06-28 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Breast Neoplasms; Psychology, Social
Keywords: Breast cancer; Latinas; Peer support counselor; Spanish speaking; Community based
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peer Support Program (Experimental): Nuevo Amanecer is the peer support program. Participants receive the peer support program as soon as possible after randomization.
  Interventions: Behavioral: Peer Support Program
- Wait-list Control (No Intervention): Waits six months, and at the end of the six months is offered the option of participating in the peer support program.

INTERVENTIONS:
Behavioral: Peer Support Program — * Work with a trained counselor who is a breast cancer survivor
  * Meet 8 times in-person over the 8 week program with the counselor
  * Counselor helps participant develop a personalized support program to help her improve her quality of life
  * Receives information on breast cancer, its treatments, and stress management
  Other Names: Nuevo Amanecer (A New Dawn)
  Arms: Peer Support Program

SUMMARY:
The purpose of this study is to test whether a new program Nuevo Amanecer (A New Dawn), improves the quality of life of Latinas diagnosed with breast cancer. Trained Latina counselors who have had breast cancer provide support to recently diagnosed women. The investigators call these counselors peer support counselors.

DETAILED DESCRIPTION:
This study will assess the effectiveness of a cognitive-behavioral stress management (CBSM) intervention for newly diagnosed Latina breast cancer patients. In our prior work, the investigators established the appropriate content of the intervention, the need for early intervention, and the value of culturally competent peer support. In this study the investigators will adapt an evidence-based CBSM intervention designed to meet these needs. This study will use a randomized controlled trial (RCT) design with a wait-listed usual care control group to adapt the intervention and test its effectiveness in improving breast cancer specific quality-of-life, and decreasing anxiety and breast cancer specific distress. The new, adapted intervention will be called "Nuevo Amanecer" (A New Dawn).

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as Latina
* Diagnosed with Stage 0, I, II, or III in the prior month
* Primarily Spanish-speaking, or Spanish monolingual
* Aged 18 or older
* Diagnosed in Alameda, Contra Costa, San Mateo, San Francisco or Santa Clara counties, California.

Exclusion Criteria:

* Previous cancer diagnosis except for non-melanoma skin cancer
* Terminal illness
* Stage IV breast cancer (distant metastasis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Gregorich, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Multiple Locations, California, United States

REFERENCES:
- [Derived] Bonilla J, Alhomsi A, Santoyo-Olsson J, Stewart AL, Ortiz C, Samayoa C, Torres-Nguyen A, Palomino H, Coleman V, Urias A, Gonzalez N, Cervantes SA, Duron Y, Napoles AM. Sharing research results with Latina breast cancer survivors who participated in a community-engaged behavioral RCT study: a descriptive cross-sectional survey study. Trials. 2022 Jan 8;23(1):25. doi: 10.1186/s13063-021-05945-8. PMID 34998436
- [Derived] Chacon L, Santoyo-Olsson J, Samayoa C, Alhomsi A, Stewart AL, Ortiz C, Escalera C, Napoles AM. Self-Efficacy for Coping with Breast Cancer Treatment Among Spanish-Speaking Latinas. Health Equity. 2021 Apr 26;5(1):245-252. doi: 10.1089/heq.2020.0152. eCollection 2021. PMID 33937611
- [Derived] Bonilla J, Escalera C, Santoyo-Olsson J, Samayoa C, Ortiz C, Stewart AL, Napoles AM. The importance of patient engagement to quality of breast cancer care and health-related quality of life: a cross-sectional study among Latina breast cancer survivors in rural and urban communities. BMC Womens Health. 2021 Feb 9;21(1):59. doi: 10.1186/s12905-021-01200-z. PMID 33563263
- [Derived] Napoles AM, Santoyo-Olsson J, Stewart AL, Ortiz C, Garcia-Jimenez M. Evaluating the Implementation of a Translational Peer-Delivered Stress Management Program for Spanish-Speaking Latina Breast Cancer Survivors. J Cancer Educ. 2018 Aug;33(4):875-884. doi: 10.1007/s13187-017-1202-y. PMID 28275966
- [Derived] Napoles AM, Ortiz C, Santoyo-Olsson J, Stewart AL, Gregorich S, Lee HE, Duron Y, McGuire P, Luce J. Nuevo Amanecer: results of a randomized controlled trial of a community-based, peer-delivered stress management intervention to improve quality of life in Latinas with breast cancer. Am J Public Health. 2015 Jul;105 Suppl 3(Suppl 3):e55-63. doi: 10.2105/AJPH.2015.302598. Epub 2015 Apr 23. PMID 25905829
- [Derived] Napoles AM, Santoyo-Olsson J, Ortiz C, Gregorich S, Lee HE, Duron Y, Graves K, Luce JA, McGuire P, Diaz-Mendez M, Stewart AL. Randomized controlled trial of Nuevo Amanecer: a peer-delivered stress management intervention for Spanish-speaking Latinas with breast cancer. Clin Trials. 2014 Apr;11(2):230-8. doi: 10.1177/1740774514521906. Epub 2014 Feb 26. PMID 24577971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from February 2011 through November 2013 via flyers and word of mouth at clinics in five Northern California counties by community recruiters.
Groups:
- Nuevo Amanecer Peer Support Program: Nuevo Amanecer is a cognitive-behavioral stress management program delivered by peers (Spanish-speaking Latinas who have had breast cancer) designed to address the first year of survivorship.
  Peer Support Program:
  * Work with a trained counselor who is a breast cancer survivor
  * Meet 8 times in-person over the 8 week program with the counselor
  * Counselor helps participant develop a personalized support program to help her improve her quality of life
  * Receives information on breast cancer, its treatments, stress management, and cognitive refraining.
Period: Baseline Assessment
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Started | 76 | 75
Completed | 76 (These 76 completed the baseline assessment and continued in the study.) | 75 (These 75 completed the baseline assessment and continued in the study.)
Not Completed | 0 | 0
Period: 3 Month Assessment
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Started | 76 | 75
Completed | 70 (These 70 completed the 3 month assessment and continued in the study.) | 74 (These 74 completed the 3 month assessment and continued in the study.)
Not Completed | 6 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Refused to complete | 4 | 0
Period: 6 Month Assessment
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Started | 76 (All 76 people were contacted at 6 months;1 person returned and 5 did not return to study at 6 months) | 74
Completed | 71 (These 71 completed the 6 month assessment and completed the study.) | 73 (These 73 completed the 6 month assessment and completed the study.)
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Refused to complete | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 66 | 70 | 136
  >=65 years | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (11.9) | 50.2 (9.9) | 50.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 75 | 151
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 76 | 75 | 151
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 76 | 75 | 151
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 76 | 75 | 151
Educational attainment [Number; unit: participants]
  Less than 6th grade | 50 | 50 | 100
  6th grade to less than high school | 15 | 12 | 27
  High school graduate | 11 | 13 | 24
Health insurance [Number; unit: participants]
  Any private | 11 | 10 | 21
  Public insurance only | 62 | 56 | 118
  None | 3 | 2 | 5
  Missing data | 0 | 7 | 7
Breast cancer [Number; unit: participants]
  Ductal Carcinoma In Situ (DCIS) | 20 | 20 | 40
  Invasive | 56 | 55 | 111
Stage [Number; unit: participants] — Stage 0-Carcinoma in situ;
  Stage I, Stage II, and Stage III-Higher numbers indicate more extensive disease: Larger tumor size and/or spread of the cancer beyond the organ in which it first developed to nearby lymph nodes and/or tissues or organs adjacent to the location of the primary tumor
  participants
    0 (in situ) | 20 | 20 | 40
    I (1) | 12 | 11 | 23
    II (2) | 31 | 26 | 57
    III (3) | 13 | 18 | 31
Surgery [Number; unit: participants]
  Breast conserving | 43 | 41 | 84
  Mastectomy | 33 | 34 | 67
Adjuvant treatment [Number; unit: participants]
  Both chemotherapy and radiation | 33 | 27 | 60
  Only radiation | 18 | 24 | 42
  Only chemotherapy | 14 | 11 | 25
  No treatment | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Physical Well-being a Subcale of the Functional Assessment of Cancer Therapy-Breast Quality of Life Instrument (FACT-B)
Description: FACT-B was used as the breast cancer-specific quality-of-life measure. FACT-B consists of 5 subscale scores pertaining to 4 well-being dimensions (physical, social-family, emotional, functional) and additional breast cancer concerns. A total overall score is the sum of all subscales. Response options were 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.
  Psychometric analysis in our Spanish-speaking Latina sample resulted in modifications to FACT-B: physical well-being subscale. Of 7 items, 1 was dropped because it was conceptually different from other items on that scale. Modified subscale was scored by summing items. Possible score ranges for physical well-being were 0-24. Higher scores indicated greater well-being.
Time Frame: Baseline and 6 month assessment
Population: Using intention-to-treat analyses, used repeated-measures linear regression models to estimate the intervention effects on outcomes. Likelihood-based model estimation assumed outcome responses were missing at random.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Number analyzed (Participants) | 76 | 75
units on a scale
  Baseline | 15.29 (5.78) | 16.76 (5.02)
  6 month | 19.44 (4.26) | 18.44 (4.58)
Statistical Analysis 1: Comparison: Nuevo Amanecer Peer Support Program vs Wait-list Control; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis — P-value represents the significance of the time by treatment group interaction from the repeated-measures linear regression model. For consistency with the manuscript, we report here the absolute means and standard deviations

2. Secondary Outcome: Anxiety a Subscale of the Brief Symptom Inventory (BSI)
Description: BSI was used to measure general symptoms of distress. BSI consists of 3 scale scores pertaining to general symptoms of distress (anxiety, depression, somatization). Response options were 0=not at all, 1=a little bit, 2=moderately, 3=quite a bit, and 4=extremely. Scores were the mean of nonmissing items. Possible score ranges for anxiety were 0-4. Higher scores indicated more distress.
Time Frame: Baseline and 6 month assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Number analyzed (Participants) | 76 | 75
units on a scale
  Baseline | 0.93 (0.84) | 1.01 (0.88)
  6 month | 0.39 (0.53) | 0.58 (0.76)
Statistical Analysis 1: Comparison: Nuevo Amanecer Peer Support Program vs Wait-list Control; Test type: Superiority or Other; p = .465, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Social/Family Well-being a Subcale of the Functional Assessment of Cancer Therapy-Breast Quality of Life Instrument (FACT-B)
Description: FACT-B was used as the breast cancer-specific quality-of-life measure. FACT-B consists of 5 subscale scores pertaining to 4 well-being dimensions (physical, social-family, emotional, functional) and additional breast cancer concerns. A total overall score is the sum of all subscales. Response options were 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.
  Psychometric analysis in our Spanish-speaking Latina sample resulted in modifications to FACT-B: social/family well-being subscale. Of 7 items, 2 were dropped because the items were conditional on having a partner (resulting in lots of missing data). Modified subscale was scored by summing items. Possible score ranges for social/family well-being were 0-20. Higher scores indicated greater well-being.
Time Frame: Baseline and 6 month assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Number analyzed (Participants) | 76 | 75
units on a scale
  Baseline | 13.67 (4.42) | 12.66 (4.25)
  6 month | 13.72 (4.81) | 14.47 (3.81)
Statistical Analysis 1: Comparison: Nuevo Amanecer Peer Support Program vs Wait-list Control; Test type: Superiority or Other; p = .025, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

4. Primary Outcome: Emotional Well-being a Subscale of the Functional Assessment of Cancer Therapy-Breast Quality of Life Instrument (FACT-B)
Description: FACT-B was used as the breast cancer-specific quality-of-life measure. FACT-B consists of 5 subscale scores pertaining to 4 well-being dimensions (physical, social-family, emotional, functional) and additional breast cancer concerns. A total overall score is the sum of all subscales. Response options were 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.
  Psychometric analysis in our Spanish-speaking Latina sample resulted in modifications to FACT-B: emotional well-being subscale. Of 6 items, 1 was dropped because of low item-scale correlations and it was conceptually different from the other items on that scale (only positively worded item on the scale). Modified subscale was scored by summing items. Possible score ranges for emotional well-being were 0-20. Higher scores indicated greater well-being.
Time Frame: Baseline and 6 month assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Number analyzed (Participants) | 76 | 75
units on a scale
  Baseline | 12.07 (4.91) | 12.86 (5.14)
  6 month | 16.39 (3.30) | 14.89 (3.95)
Statistical Analysis 1: Comparison: Nuevo Amanecer Peer Support Program vs Wait-list Control; Test type: Superiority or Other; p = .004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

5. Primary Outcome: Breast Cancer Concerns a Subscale of the Functional Assessment of Cancer Therapy-Breast Quality of Life Instrument (FACT-B)
Description: FACT-B was used as the breast cancer-specific quality-of-life measure. FACT-B consists of 5 subscale scores pertaining to 4 well-being dimensions (physical, social-family, emotional, functional) and additional breast cancer concerns. A total overall score is the sum of all subscales. Response options were 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.
  Psychometric analysis in our Spanish-speaking Latina sample resulted in modifications to FACT-B: breast cancer concerns subscale. Of 7 items, 2 were dropped because of low item-scale correlations and were conceptually different from the other items on that scale. Modified subscale was scored by summing items. Possible score ranges for emotional well-being were 0-28. Higher scores indicated greater well-being.
Time Frame: Baseline and 6 month assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Number analyzed (Participants) | 76 | 75
units on a scale
  Baseline | 16.52 (5.43) | 17.33 (5.08)
  6 month | 21.31 (3.83) | 19.92 (5.22)
Statistical Analysis 1: Comparison: Nuevo Amanecer Peer Support Program vs Wait-list Control; Test type: Superiority or Other; p = .013, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

6. Primary Outcome: Enjoyment of Life a Subscale of the Functional Assessment of Cancer Therapy-Breast Quality of Life Instrument (FACT-B)
Description: FACT-B was used as the breast cancer-specific quality-of-life measure. FACT-B consists of 5 subscale scores pertaining to 4 well-being dimensions (physical, social-family, emotional, functional) and additional breast cancer concerns. A total overall score is the sum of all subscales. Response options were 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.
  Psychometric analysis in our Spanish-speaking Latina sample resulted in modifications to FACT-B: functional well-being subscale. Of 7 items, 3 were dropped because items were conceptually different and did not converge psychometrically with the other items on that scale; the remaining 4 items were specific to enjoyment of life, thus we renamed the subscale to "Enjoyment of Life". Modified subscale was scored by summing items. Possible score ranges for enjoyment of life were 0-16. Higher scores indicated greater well-being.
Time Frame: Baseline and 6 month assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Number analyzed (Participants) | 76 | 75
units on a scale
  Baseline | 8.92 (3.80) | 9.22 (3.43)
  6 month | 9.79 (3.39) | 9.30 (3.06)
Statistical Analysis 1: Comparison: Nuevo Amanecer Peer Support Program vs Wait-list Control; Test type: Superiority or Other; p = .267, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

7. Primary Outcome: Total Score of the Functional Assessment of Cancer Therapy-Breast Quality of Life Instrument (FACT-B)
Description: FACT-B was used as the breast cancer-specific quality-of-life measure. FACT-B consists of 5 subscale scores pertaining to 4 well-being dimensions (physical, social-family, emotional, functional) and additional breast cancer concerns. A total overall score is the sum of all subscales. Response options were 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.
  Psychometric analysis in our Spanish-speaking Latina sample resulted in modifications to each of the FACT-B subscale. The total overall score is based on the sum of modified subscales (see above primary outcomes for modifications to subscales). Possible score ranges for the total overall score were 0-108. Higher scores indicated greater well-being.
Time Frame: Baseline and 6 month assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Number analyzed (Participants) | 76 | 75
units on a scale
  Baseline | 66.46 (16.92) | 68.83 (15.33)
  6 month | 80.64 (13.64) | 77.02 (15.62)
Statistical Analysis 1: Comparison: Nuevo Amanecer Peer Support Program vs Wait-list Control; Test type: Superiority or Other; p = .030, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Depression a Subscale of the Brief Symptom Inventory (BSI)
Description: BSI was used to measure general symptoms of distress. BSI consists of 3 scale scores pertaining to general symptoms of distress (anxiety, depression, somatization). Response options were 0=not at all, 1=a little bit, 2=moderately, 3=quite a bit, and 4=extremely. Scores were the mean of nonmissing items. Possible score ranges for depression were 0-4. Higher scores indicated more distress.
Time Frame: Baseline and 6 month assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Number analyzed (Participants) | 76 | 75
units on a scale
  Baseline | 0.93 (0.84) | 0.75 (0.76)
  6 month | 0.38 (0.48) | 0.46 (0.62)
Statistical Analysis 1: Comparison: Nuevo Amanecer Peer Support Program vs Wait-list Control; Test type: Superiority or Other; p = .045, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Somatization a Subscale of the Brief Symptom Inventory (BSI)
Description: BSI was used to measure general symptoms of distress. BSI consists of 3 scale scores pertaining to general symptoms of distress (anxiety, depression, somatization). Response options were 0=not at all, 1=a little bit, 2=moderately, 3=quite a bit, and 4=extremely. Scores were the mean of nonmissing items. Possible score ranges for somatization were 0-4. Higher scores indicated more distress.
Time Frame: Baseline and 6 month assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Number analyzed (Participants) | 76 | 75
units on a scale
  Baseline | 0.93 (0.78) | 0.75 (0.59)
  6 month | 0.52 (0.51) | 0.66 (0.60)
Statistical Analysis 1: Comparison: Nuevo Amanecer Peer Support Program vs Wait-list Control; Test type: Superiority or Other; p = .005, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Breast Cancer-Specific Distress of the Intrusive Thoughts Scale
Description: Breast cancer-specific distress was measured with the 7 item Intrusive Thoughts Scale (anchored to the breast cancer experience), a subscale of the revised Impact of Event Scale (RIES). Response options were 0=not at all, 1=rarely, 2=sometimes, and 3=often. Using the published scoring algorithm, items were summed after recoding responses to 0, 1, 3, and 5. Possible score ranges were 0-35. Higher scores indicate greater distress.
Time Frame: Baseline and 6 month assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Number analyzed (Participants) | 76 | 75
units on a scale
  Baseline | 7.96 (8.46) | 8.65 (8.91)
  6 month | 3.87 (5.79) | 6.27 (8.42)
Statistical Analysis 1: Comparison: Nuevo Amanecer Peer Support Program vs Wait-list Control; Test type: Superiority or Other; p = .226, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Nuevo Amanecer Peer Support Program | Wait-list Control
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 0/76 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No